CLINICAL TRIAL: NCT01593813
Title: Repair or Not Repair Pronator Quadratus in the Volar Plating of Distal Radial Fracture-Are Functional Outcomes Differ ?
Brief Title: Repair or Not Repair Pronator Quadratus in the Volar Plating of Distal Radial Fracture Are Functional Outcomes Differ ?
Acronym: PQ
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Principal Investigator, National Taiwan University Hospital, Zheng Ren Dong, National Taiwan University Hospital
Other Study IDs: PQ repair
Record Dates: First submitted 2012-05-04; First posted 2012-05-08 (Estimated); Last update posted 2012-05-08 (Estimated); Status verified 2012-05

CONDITIONS: Distal Radius Fracture
Keywords: Pronator quadratus; distal radius fracture; volar plating
MeSH Terms: conditions — Wrist Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The theoretical benefits of the repair of the pronator quadratus include flexor tendon protection, remain of the normal pronation-supination range of motion (ROM) and strength, and keeping the stable DRUJ.

Repair or not repair pronator quadratus in the volar plating of distal radial fracture-Are functional outcomes differ?

DETAILED DESCRIPTION:
In the operation of distal radial fractures, the volar plating techniques become popular. During the surgical approach, the pronator quadratus (PQ) muscle needs split or full-thickness strip to exposure the fracture site and facilitate the instrumentation of the plate. Generally, the PQ would be repaired. Sometimes, the PQ is damaged by the fracture fragment so severely that it is difficult to repair the PQ. However, there is few reviews paper to discuss the consequence of the unrepaired or repaired PQ and the AAOS guideline1 of the treatment of distal radial fracture in 2009 did not even list the management of the PQ. The function of the PQ includes pronation and stability of the distal radial-ulnar joint (DRUJ). According to the study, the elimination of PQ function will cause a significant decrease in pronation torque, which is supposed to affect the function of the wrist in the daily life. The theoretical benefits of the repair of the pronator quadratus include flexor tendon protection3,4, remain of the normal pronation-supination range of motion (ROM) and strength, and keeping the stable DRUJ.

ELIGIBILITY:
Inclusion Criteria:

* ≧ 20 or ≦ 80-years-old adult patients
* Cooperative to evaluation
* Distal radial fracture, fresh, single fracture
* Volar plating

Exclusion Criteria:

* < 20 or > 80-years-old patients
* Uncooperative adult, such as dementia
* Old fracture, more than 1 Week
* Multiple fractures
* Pathological fracture
* Surgery other then volar plating

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patient with distal radius fracture
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2012-05; Primary Completion 2013-03 (Estimated); Study Completion 2013-03 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Jui-sheng Sun, PHD, Study Chair — Department of Orthopedics of NTUH